CLINICAL TRIAL: NCT05130151
Title: Using Mobile Technology to Prevent HIV and Related Youth Health Problems: Sexual Health, Mental Health and Substance Use in Southwest Uganda
Brief Title: Using Mobile Technology to Prevent HIV and Related Youth Health Problems
Acronym: YouthHealth
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: U.S. Department of HHS OHRP issued an FWA restriction on NYSPI research that included a pause of human subjects research as of June 23, 2023. This study will resume recruitment after OHRP has approved the resumption of research.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Washington University School of Medicine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Philip Kreniske, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8183; K01MH122319 (NIH)
Record Dates: First submitted 2021-11-01; First posted 2021-11-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Adolescents (N = 200) will be randomized into two arms - 100 into the adapted mobile phone-based intervention arm, and 100 into standard education provided in schools.
Who Masked: Participant, Care Provider
Masking Description: Participants and providers are the parties involved in the clinical trial who are prevented from having knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will receive the mobile phone-based intervention.
  Interventions: Behavioral: Youth Health SMS
- Standard of care (No Intervention): Participants in this arm will receive only standard of care.

INTERVENTIONS:
Behavioral: Youth Health SMS — The intervention is comprised of an automated two-way text messaging and interactive voice recognition service that provides sexual reproductive health (SRH) and HIV prevention information. The proposed intervention will add PrEP information and mental health and alcohol use screeners to the platform with the goal of promoting linkage to HIV clinics and to phone-based mental health counseling for symptomatic participants.
  Arms: Intervention

SUMMARY:
Since the start of this study I have moved from NYSPI to City University of New York. The study is currently paused.

The goal of the project is to find out how the investigators can use mobile phones to prevent HIV and address related health problems such as sexual health and mental health among adolescents. The investigators will evaluate and adapt an existing text-message and interactive voice recognition (IVR) system. IVR is Interactive voice response is a technology that allows humans to interact with a computer-operated phone system through the use of voice and DTMF tones input via a keypad.

The system was designed by FHI 360 (note FHI 360 is the name of the non-profit not an acronym). FHI 360 is an international nonprofit working to improve the health and well-being of people in the United States and around the world. FHI 360 staffs more than 4,000 professionals who work in more than 60 countries. Examples of the existing content is available (https://m4rh.fhi360.org/?page_id=191) and we have a letter of support from FHI 360, included in my funded grant proposal, stating we may use and modify this content as needed. As noted below anyone can access this content by dialing #161 when in Uganda. FHI 360 sexual reproductive health information is currently available across Uganda for free and can be accessed in by dialing #161.

The proposed research comprises two phases. Phase 1 involves two steps, (A) "theater pretesting" (includes brief interviews) (B) focus groups (or more detailed interviews depending on COVID-19 guidelines and described in detail below) that will involve asking adolescents to discuss new messages that would provide basic information about pre-exposure prophylaxis (PrEP) as well as, a set of questions about mental health, and alcohol use. We will conduct focus groups with these adolescents and elicit responses to improve the acceptability of the messages (described in detail below).

We will then modify any content as needed and conduct Phase 2 which involves (A) randomized control trial and (B) qualitative key informant interviews. Adolescents (N=200) will be randomly assigned to either the mobile phone-based intervention or to standard of care. Through this approach we will evaluate our adaptation of FHI 360's existing text message and interactive voice recognition (IVR). The adaptation will include PrEP information as well as specific mental health and hazardous alcohol use screens, promote HIV prevention for all adolescents, and support linkage to behavioral health counselors for symptomatic adolescents.

DETAILED DESCRIPTION:
Background This study will result in the development of one of the first mobile phone-based interventions for adolescents in East Africa that begins to address sexual health, mental health, and alcohol use. Adolescence is a developmental period associated with the increased importance of peers, increased technology use, increased mobility, initiation of sex, emergence of mental health disorders (if at risk), and initiation of alcohol use. Thus, the initial step of screening and linking adolescents with mental health or alcohol use problems to counselors, may help address these factors and also reduce the risk for HIV infection. Further, PrEP has only recently been made available to adolescents in Uganda and is not currently included in the existing FHI 360 #161 system. As described by the CDC, PrEP is a way for people who do not have HIV but who are at very high risk of getting HIV to prevent HIV infection by taking a pill every day. Studies have shown that PrEP reduces the risk of getting HIV from sex by about 99% when taken daily. Adolescents today rely heavily on mobile phones for information and services, thus the investigators believe the proposed intervention could be applied and adapted across the region, and potentially in other under-resourced settings.

Aim 1: To adapt an evidence-based mobile phone-delivered sexual health program, to include PrEP information and deliver mental health and alcohol use assessments with the goal of increasing screening and referral, as well as linkage to school-based counselors for adolescents at HIV risk.

Aim 2: Evaluate through a pilot RCT (N=200 adolescents, 15-19 years) intervention (a) acceptability and feasibility, and (b) impact on uptake of HIV prevention strategies, as well as screening and linkage to mental health and alcohol use school-based counselors.

For aim 2 the investigators hypothesize that the intervention group will uptake HIV testing and a greater rate than the control group.

Procedures There will be two phases to the study. The first will last approximately three months and include 24 subjects (15-19 years). The second phase will include 200 subjects (15-19 years) with a five week intervention and a follow-up survey within six monthhs.

The professional networks of Dr. Fred Ssewamala (K01 advisor) will be used to recruit schools with potential participants. Dr. Ssewamala is the director of the International Center for Child Health and Development (ICHAD) at the Washington University in St. Louis (WUSTL) School of Medicine. ICHAD and Ssewamala have multiple NIH-funded studies among the target population for the current study and existing relationships with local secondary schools and community leaders. The study Project Director, a masters student at WUSTL and Ugandan national, will contact ICHAD partnered schools and local community leaders using the attached text adapted from prior studies in the region (see Recruitment Materials). The Project Director and Research Assistant will work primarily out of the ICHAD offices in Masaka Uganda.

The existing intervention, designed by the international health organization FHI 360 and regional technology partner Viamo, with Ugandan offices in Kampala, works through SMS or by calling a designated short code, which in Uganda is *161. The system then automatically responds with a menu of choices for accessing HIV prevention and contraceptive information, as well as HIV clinic locations. To select an option, the user replies with an SMS using a keyword or code from the provided menu. For example, "press 5 for HIV prevention" (see phone number in Facilities for access to further examples). The system then provides an auto response to the user.

Our intervention, again working with regional tech-partner Viamo, will add to the current HIV prevention menu, information on PrEP, such as "PrEP, is a way to help prevent HIV by taking a pill every day," Texting or calling this platform is free in Uganda and across East Africa due to agreements between FHI360, the tech company Viamo, and regional phone networks. All messages will be provided in English or Luganda.

The Project Director and the Research Staff will be the primary research staff to interact with participants. If needed Dr Ssewamala or PI Kreniske would assist. Depending on COVID-19 guidelines Dr. Kreniske may have the opportunity to directly interact with study participants. For example, if possible, Kreniske would travel to Uganda at to observe the Phase 1 or Phase 2 focus groups or interviews that could be conducted in English or Luganda depending on the participants preferences. If needed, as a backup Kreniske would also assist in conducting interviews or focus groups.

If more adolescents express interest in participating in Phase I of the study than are needed the investigators will keep their contact information in a secure locked filing cabinet or encrypted laptop so that the investigators can reach them for potential participation in Phase II. If more adolescents than are needed express interest in Phase II the investigators will inform them that recruitment has concluded and thank them for their interest.

Phase 1 involves two steps, (A) "theater pretesting" with daily brief individual interviews (B) focus groups. Participants will be explicitly informed by the Project Director or Research Assistant and via the consent form, that they are entitled to refrain from answering any questions that arise during the interview or focus group which they do not wish to answer. All interviews and focus groups will be audio recorded. Audio files will be immediately moved to the Project Director's password protected, encrypted computer and deleted after 1 year. Consistent with ongoing ICHAD research in the region, compensation for adolescent participation will include US $7.33 in Uganda shillings in cash which will be administered to the participant by the Project Director or Research Assistant at the completion of interviews. The Project Director or Research Assistant have completed necessary Collaborative Institutional Training Initiative (CITI) courses including Good Clinical Practice (GCP) and Human Subjects Protection SBR with minors.

Theater pretesting involves developing the messages and concepts of an intervention and exploring them with intended audiences, in this study - young people (15-19 years) (Table 6). During theater pretesting 24 (12 men, 12 women) potentially eligible participants, referred by members of local schools or local council members, will be prompted to view or listen to and interact with the adapted mobile phone intervention messages and menus. Each day over a 1-week period adolescents will be prompted to interact with a different component of the intervention generally requiring them to listen to about 5-7 messages or respond to 5-7 questions on the following topics (e.g. HIV prevention, HIV clinic locator, mental health screen using The Patient Health Questionnaire (PHQ-9), The Generalized Anxiety Disorder Questionnaire (GAD-7) and alcohol use screen using the Alcohol Consumption Questions-C (AUDIT-C). To ensure the investigators maintain confidentiality only adolescents who own their phones will be recruited to the study. Text messages pop-up on the screen with the notification 1 new message. However, only a person who has the password to the phone can access the message.

Viamo's IVR-text-messaging system will be programmed to score responses to these measures in the following way: If the respondents score 0 the system will respond with an auto message thanking them for their responses. If respondents score a 1 or greater on the PHQ-2 + i9 or GAD-7 they will then be given the full measures. In addition, the investigators will contact the StrongMinds counselors and local agencies and follow established ICHAD procedures if any respondent endorses the following suicide question "Thoughts that you want to kill yourself, or have you attempted suicide?".

Following this interaction participants will be contacted by our study coordinator or research assistant and asked a series of brief questions to assess the intervention components through an audio recorded phone call: (1) content (e.g. themes, materials, role-play vignettes); (2) delivery; and (3) activities that may not be addressed to enhance the intervention relevance. The investigators anticipate interacting with the platform and the subsequent rapid interview will require a total of 10 minutes per day. At the end of the week to assess acceptability, all 24 adolescents will be asked to complete a 12-item survey to evaluate acceptability. This measure will be administered over the phone by the Project Director or Research Assistant. To further evaluate feasibility, the investigators will use measures previously used by FHI 360, including number of messages viewed, type of messages viewed and number of times the service locator was used. The investigators will also measure number of attempted and completed mental health and alcohol screens, and the use of counselor referrals. As described below, the investigators will refer to StrongMinds, a non-governmental organization who currently provide free mobile phone-based mental health counseling in Uganda. Consistent with previous work, all messages to the system will be tracked through electronic logging of message source (mobile phone number), type of information (e.g. HIV prevention) and date and time of the message.

The investigators will then conduct 4 focus groups with 5-6 participants each. The purpose of the focus groups, approximately 45-minute each, is to gather preliminary understanding of feasibility and acceptability and determine if modifications are needed. Currently, Uganda is allowing people to gather in small groups under national mitigation strategies for research. Depending on the COVID-19 guidelines at the time of the data collection the investigators are prepared to hold in person interviews with COVID-19 precautions including social distancing, required masks, and an outdoor meeting space or to conduct the groups over the phone if the COVID-19 guidelines change. Areas of focus will include (a) the acceptability of the new PrEP information, (b) Adolescents feedback on clinic referral message content, (c) preferences for daily, weekly or no unsolicited messages, and (d) identifying technical issues. All adolescents will also complete a brief acceptability measure that was used previously for adolescents in Uganda. Responses to these questions will be used to facilitate adapting the intervention to the adolescents 15-19 in Uganda.

In Phase 2, prior to the full randomized controlled pilot trial the investigators will soft launch the adapted intervention with a group of 10 adolescents over a 1-month period. A soft launch is often used in product development to identify any technical issues prior to a full rollout or trial. The investigators will also employ a paired down version of the pre-post assessments and questions of feasibility and acceptability with this group. This process will allow us to correct any issues with the system prior to conducting the full trial. The investigators will then conduct a pilot trial of the adapted mobile phone-based intervention over 9 months. Adolescents (N = 200) will be randomized into two arms - 100 into the adapted mobile phone-based intervention arm, and 100 into standard education provided in schools.

Standard of care. Two curricula are delivered in all secondary schools in Uganda: Life Planning Skills and Adolescent Sexual Reproductive Health (ASRH). This is considered usual care in our study, and all enrolled participants, both in control and treatment conditions, will be exposed to these curricula. In the curricula, the content related to HIV and sexual risk-taking behaviors includes delaying sex; using condoms and contraception; and preventing substance abuse. This curriculum also includes education on gender equality and importance of delayed marriage. The content is primarily delivered via class lectures. The ASRH content is dispersed across a range of academic subjects in secondary schools. In each class, students receive information about sexual activity, HIV prevention, and gender studies relevant to that subject. Teachers and students all receive a sex and health education handbook

Following the intervention the investigators will conduct 30 key informant interviews (KII) with adolescents in the intervention arm. SRH and PrEP information is not currently included in the Ugandan standard curricula, nor are mental health or substance use assessments.

The investigators plan to use a simple text reminder such as "Reach out and contact *161 for your weekly check-in!". The weekly mobile check-in will require about 10-minutes of participants time per week.

Starting at baseline and each subsequent week (1 months total) participants will receive a text message prompting them to interact with one menu. These menus include Current HIV Prevention Strategies (including PrEP), SRH Clinic Locator, Depression Screen (PHQ-9), Anxiety Disorder Screen (GAD-7), Alcohol Use Disorders Screen (AUDIT). As our primary outcome is HIV testing adolescents will be prompted to interact with the Current HIV Prevention Strategies (including PrEP) and SRH Clinic Locator in the first 2 weeks and the final 2 weeks of the study.

In addition, participants will be asked to complete survey responses at baseline, with 6 months post intervention later. Table 1 included below in the "assessment instrument" section lists the full survey battery.

Finally, immediately post-intervention the investigators will conduct 30 KII with participants in the intervention group. Feasibility questions will be asked in relation to texting barriers.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents (aged 15-19 years): Self-report during enrollment and confirmed by school personnel or local community leader.
2. Residing in the greater Masaka region in southern Uganda: Self-report during enrollment and confirmed by school personnel or local community leader.
3. Own a mobile phone: Self-report during enrollment and confirmed visually by project director or research assistant.
4. People who have the cognitive capacity to consent: A potential participant will be included if the researcher conducting the consent process determines that the potential participant has the cognitive capacity to consent. This will be determined by through the review of the consent forms.
5. For Phase II, did not participate. In Phase I: Review of study records.

Exclusion Criteria:

1. People who are not aged 15-19 years: Self-report during enrollment and confirmed by school personnel or local community leader.
2. People who do not reside in the greater Masaka region in southern Uganda: Self-report during enrollment and confirmed by school personnel or local community leader.
3. People who do not own a mobile phone: Self-report during enrollment and confirmed visually by project director or research assistant.
4. People who do not have the cognitive capacity to consent: A potential participant will be excluded if the researcher conducting the consent process determines that the potential participant has a mental deficit or does not have the cognitive capacity to understand the consent process and proposed research.
5. Participants in phase 1 will be excluded from phase 2: Review of study records

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
HIV-AIDS Test | 6 month
  Self-report and verified at local clinic number of HIV Tests

SECONDARY OUTCOMES:
Depression | 6 month
  Pre-Post Scores of Depression as measured by the The Patient Health Questionnaire (PHQ-9). The Patient Health Questionnaire (PHQ-9)(Kroenke K & Spitzer RL, 2001) - a standardized 9-item self-report instrument - was used to assess depression. Participants rate the frequency of their symptoms over the past 2 weeks. Items are rated on a 4-point scale from 0 (not at all) to 3 (nearly every day) and scale scores range from 0 to 27. PHQ-9 scores of 5-9, represent minimal to mild depression, and 10-20 represent moderate to severe depression. As recommended, PHQ-9 scores ≥ 10 were considered indicative of screening positively for clinically significant depressive symptoms (Kroenke K & Spitzer RL, 2001). The PHQ-9 has good test-retest reliability and validity. A score equal to or greater than 10 has a sensitivity of 88% and a specificity of 88% for major depression (Kroenke K & Spitzer RL, 2001).
Alcohol Use | 6 month
  Pre-Post Alcohol use scores Alcohol Consumption Questions (AUDIT or AUDIT-C). The AUDIT-C (Bohn et al., 1995) is a 3-item screener excerpted from the full standardized 10-item AUDIT tool to assess hazardous alcohol consumption. Items are scored on a 5-point scale for a possible score of 0 to 12. The higher the score, the higher the risk of hazardous alcohol consumption. An AUDIT-C score of 4 or greater in men, and 3 or greater in women is considered positive for hazardous alcohol consumption (Bohn et al., 1995)
PrEP Use | 6 month
  Pre-Post PrEP Use based on self-report.
Anxiety | 6 month
  Pre-Post Scores of The Generalized Anxiety Disorder Questionnaire (GAD-7). The GAD-7 is a standardized instrument that asks participants to rate their symptoms over the past two weeks on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Overall scores for the GAD-7 range from 0 to 21. At a cut-point of 10 (indicative of clinically significant symptoms), the sensitivity and specificity of the scale equals 89% and 82% respectively. The GAD-7 has a Cronbach's alpha of .92, indicating good internal consistency with an intra-class correlation of .83, indicating good procedural validity (Spitzer et al., 2006).
Mental Health Counseling | 6 month
  Mental Health Counseling sessions self-reported.

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from the proposed application will be uploaded no more than three months after the trial has been completed. This will enable other research groups to access these de-identified data.
Supporting Information: Study Protocol, SAP
Time Frame: This will be provided no more than three months after the trial has been completed.
Access Criteria: We will upload to clinicaltrials.gov

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Olsen PS, Plourde KF, Lasway C, van Praag E. Insights From a Text Messaging-Based Sexual and Reproductive Health Information Program in Tanzania (m4RH): Retrospective Analysis. JMIR Mhealth Uhealth. 2018 Nov 1;6(11):e10190. doi: 10.2196/10190. PMID 30389651
- [Background] Bohn MJ, Babor TF, Kranzler HR. The Alcohol Use Disorders Identification Test (AUDIT): validation of a screening instrument for use in medical settings. J Stud Alcohol. 1995 Jul;56(4):423-32. doi: 10.15288/jsa.1995.56.423. PMID 7674678
- [Background] Johnson D, Juras R, Riley P, Chatterji M, Sloane P, Choi SK, Johns B. A randomized controlled trial of the impact of a family planning mHealth service on knowledge and use of contraception. Contraception. 2017 Jan;95(1):90-97. doi: 10.1016/j.contraception.2016.07.009. Epub 2016 Jul 13. PMID 27421767
- [Background] Vahdat HL, L'Engle KL, Plourde KF, Magaria L, Olawo A. There are some questions you may not ask in a clinic: providing contraception information to young people in Kenya using SMS. Int J Gynaecol Obstet. 2013 Nov;123 Suppl 1:e2-6. doi: 10.1016/j.ijgo.2013.07.009. Epub 2013 Aug 2. PMID 24012514
- [Derived] Kreniske P, Namuyaba OI, Kasumba R, Namatovu P, Ssewamala F, Wingood G, Wei Y, Ybarra ML, Oloya C, Tindyebwa C, Ntulo C, Mujune V, Chang LW, Mellins CA, Santelli JS. Mobile Phone Technology for Preventing HIV and Related Youth Health Problems, Sexual Health, Mental Health, and Substance Use Problems in Southwest Uganda (Youth Health SMS): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Dec 19;12:e49352. doi: 10.2196/49352. PMID 38113102